CLINICAL TRIAL: NCT03539107
Title: Voiding Assessment Based on Minimum Spontaneous Void of 150 mL Compared to Retrograde Fill Method After Female Pelvic Floor Reconstructive Surgery: A Randomized Controlled Trial
Brief Title: Voiding Assessment Based on Minimum Spontaneous Void of 150 mL Compared to Retrograde Fill Method After Female Pelvic Floor Reconstructive Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Popiel02
Record Dates: First submitted 2018-05-15; First posted 2018-05-29 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Urinary Incontinence; Pelvic Organ Prolapse
MeSH Terms: conditions — Urinary Incontinence; Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spontaneous void (Experimental): Subjects will not have retrograde fill of bladder, rather will be required to void 150 mL spontaneously prior to discharge.
  Interventions: Other: spontaneous void
- Retrograde bladder fill (Active Comparator): Subjects will have their bladder retrograde filled with 300mL of fluid prior to a voiding trial.
  Interventions: Procedure: Retrograde bladder fill

INTERVENTIONS:
Procedure: Retrograde bladder fill — Subjects will have their bladder retrograde filled with 300mL of fluid prior to a voiding trial.
  Arms: Retrograde bladder fill
Other: spontaneous void — Subjects will not have retrograde fill of bladder, rather will be required to void 150 mL spontaneously prior to discharge.
  Arms: Spontaneous void

SUMMARY:
This study will compare voiding assessment based on a minimum spontaneous voided volume of 150 cc with the standard retrograde fill approach in women after pelvic floor procedures.

ELIGIBILITY:
Inclusion Criteria:

* All 18-year-old or older women who undergo surgery for urinary incontinence and/or pelvic organ prolapse (POP)

Exclusion Criteria:

* Patients who require prolonged Foley catheter or suprapubic catheter

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Failure rate | Up to 2 days post op
  The percentage of subjects who did not meet the required voiding assessment criteria and needed catheterization .

SECONDARY OUTCOMES:
False pass rate | up to 30 days after discharge.
  The percentage of women who initially met the voiding assessment but returned for re-catheterization due to voiding difficulty .
Force of stream (FOS) | Up to 2 days post op.
  Patient reported force of stream (FOS) during voiding; (0 being no urination, 10 being normal strong flow).
Force of stream (FOS) | Up to 2 days post-surgery.
  Patient reported force of stream (FOS) during voiding; (0 being no urination, 10 being normal strong flow).
Patient Satisfaction Questionnaire for Voiding Assessment-method used | Up to 2 days post-surgery.
  This question asks "How satisfied were you with the method we used to evaluate how well you could urinate after our surgery?" It is measured on a continuum from 0 (very dissatisfied) to 100 (very satisfied).
Patient Satisfaction Questionnaire for Voiding Assessment-negative emotions | Up to 2 days post-surgery.
  This question asks "Did you experience any negative emotions such as fear or anxiety when we were evaluating urination after our surgery?" It is measured on a continuum from 0 (many negative emotions) to 100 (no negative emotions).
Patient Satisfaction Questionnaire for Voiding Assessment-recommend method | Up to 2 days post-surgery.
  This question asks "How likely would you be to recommend to a friend or family member, the method we used to evaluate your urination after our surgery, if they were in the same situation?" It is measured on a continuum from 0 (very unlikely) to 100 (very likely).
Patient Satisfaction Questionnaire for Voiding Assessment-convenience of method | Up to 2 days post-surgery.
  This question asks "How convenient was the method we used to evaluate your urination after our surgery (e.g. time, ease etc.)? It is measured on a continuum from 0 (very inconvenient) to 100 (very convenient).
Patient Satisfaction Questionnaire for Voiding Assessment-preferred method | Up to 2 days post-surgery.
  This question asks the patient: "If it was all up to you, which It is measured on a continuum from 0 (strongly prefer backfill before catheter) to 100 (strongly prefer no backfill before catheter removal).
Postoperative pain score | One day post-surgery.
  This outcome is measured by a 10-point visual analog scale where 0= no pain, 10=worst pain you have ever experienced.
Urinary tract infection (UTI) | Up to 30 days post surgery.
  UTI is defined as culture-proven bladder infection or, in the absence of a culture, clinical suspicion of a bladder infection that resulted in treatment.
Post-operative complications | Up to 30 days post-surgery.
  Post-operative complications assessed by medical record review.
Length of hospital stay | Up to 2 days post-surgery.
  Length of hospital stay assessed by medical record review.

CONTACTS AND LOCATIONS:
Overall Officials: Harmanli Oz, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246